CLINICAL TRIAL: NCT03234621
Title: Protective Ventilation Strategy During One-lung Ventilation: Effect on Postoperative Pulmonary Complications
Brief Title: Protective Ventilation Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Hyon Bahk, MD, PhD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JHBahk_PV
Record Dates: First submitted 2017-07-26; First posted 2017-07-31 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2017-07

CONDITIONS: One-lung Ventilation
Keywords: protective ventilation strategy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional tidal group (Experimental): provide tidal volume of 6ml/kg (predicted body weight) with positive end expiratory pressure of 5cmH2O during one-lung ventilation
  Interventions: Other: ventilator setting during one-lung ventilation
- low tidal group (Experimental): provide tidal volume of 4ml/kg (predicted body weight) with positive end expiratory pressure of 5cmH2O during one-lung ventilation
  Interventions: Other: ventilator setting during one-lung ventilation
- high tidal group (Experimental): provide tidal volume of 8ml/kg (predicted body weight) with positive end expiratory pressure of 5cmH2O during one-lung ventilation
  Interventions: Other: ventilator setting during one-lung ventilation

INTERVENTIONS:
Other: ventilator setting during one-lung ventilation — providing various tidal volumes according to the groups with constant PEEP

SUMMARY:
The purpose of this study is to find a proper ventilation strategy for one-lung ventilation to prevent postoperative pulmonary complications

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective thoracic surgery
* ASA I, II, III
* scheduled > 2 hours of surgery

Exclusion Criteria:

* denied patients
* age under 18 years
* FEV1/FVC or FEV1<70% in preoperative pulmonary function test

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
postoperative pulmonary complications | immediately after operation
  PaO2/FiO2 and/or newly appeared atelectasis, lung infiltration

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea